CLINICAL TRIAL: NCT02858557
Title: The Effect of the Mediterranean Diet and the Specific Carbohydrate Diet on Microbial Profile and Disease Outcomes in Patients With Inflammatory Bowel Diseases
Brief Title: The Effect of Diet on Microbial Profile and Disease Outcomes in Patients With Inflammatory Bowel Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0240-16-TLV
Record Dates: First submitted 2016-07-28; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Inflammatory Bowel Diseases; Crohn's Disease; Dietary Modification
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Patients will be allocated to 7 days of Mediterranean diet and then will cross over to 7 days of specific carbohydrate diet
  Interventions: Behavioral: Mediterranean diet; Behavioral: Specific Carbohydrate Diet
- Group B (Experimental): Patients will be allocated to 7 days of specific carbohydrate diet and then will cross over to 7 days of Mediterranean diet
  Interventions: Behavioral: Mediterranean diet; Behavioral: Specific Carbohydrate Diet

INTERVENTIONS:
Behavioral: Mediterranean diet — The Mediterranean diet is rich in complex carbohydrates and fibers and low in animal proteins and fats.
Behavioral: Specific Carbohydrate Diet — The specific carbohydrate diet is a dietary program popular among patients with IBD. The diet allows carbohydrate foods consisting of mono-saccharides only, and excludes di-saccharides and most polysaccharides.

SUMMARY:
This clinical study is designed to evaluate the effect of two dietary patterns, Mediterranean diet and the specific carbohydrate diet on clinical, inflammatory and microbial parameters in patients after pouch surgery and to assess the effect of a personal tailored diet, based on microbial profile, on disease outcomes and generate a predictive model for future interventions.

DETAILED DESCRIPTION:
Increasing evidence exist regarding the role of diet in the pathogenesis of inflammatory bowel diseases. One possible mechanism for the effect of diet on intestinal inflammation is modification of the gut microbial composition. However, the relationship between diet, the microbiome and intestinal inflammation is still vague.

The investigators plan to perform a crossover clinical trial. Seventy ulcerative colitis patients post restorative proctocolectomy (pouch) will be randomly allocated into two short-term (one week) dietary interventions, the Mediterranean diet and the specific carbohydrate diet, to assess which diet has the required influence (i.e. increased diversity, decrease in specific pathobionts and increase in "anti-inflammatory" taxa) on the gut microbiome of each participant. Based on this assessment, each participant will be treated by a personally-tailored diet for up to one year, during which microbial composition, clinical parameters, and quality of life will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75;
* Able and willing to sign an informed consent;
* Underwent pouch surgery because of refractory UC or Familial Adenomatous Polyposis (FAP) and have a functioning pouch.

Exclusion Criteria:

* Patients with ileostomy, stricturing disease, use of antibiotics in the month prior to inclusion, significant comorbidity that precludes the patient from participating according to the physicians' judgment, non-Hebrew readers, pregnant and lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Microbial diversity | 7 days
  Shannon α-diversity index

SECONDARY OUTCOMES:
Clinical score | 7 days
  Pouchitis Disease Activity Index (PDAI)
C-reactive protein (CRP) | 7 days
  Inflammatory marker
fecal calprotectin | 7 days
  Inflammatory marker
Quality of life | 7 days
  Inflammatory bowel diseases questionnaire (IBDQ)
Microbial composition | 7 days
  Change in the abundance of microbial taxa

CONTACTS AND LOCATIONS:
Overall Officials: Iris Dotan, MD, Principal Investigator — Head, IBD center, Department of gastroenterology and liver diseases, Tel Aviv Sourasky Medical Center
Locations (1):
- Dep. of Gastroenterology, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No